CLINICAL TRIAL: NCT06259513
Title: Feasibility of Tailoring Axillary Surgery Based on the Molecular Subtype and Nodal Burden of Breast Cancer Patients- SentiOMIT and SentiMACRO Trial
Brief Title: Omission of Axillary Surgery in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB Ref: 2023/2735
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients with omission of SLNB (Experimental): early breast cancer patients with cT1-2N0 Luminal A subtype with omission of SLNB
  Interventions: Procedure: omission of SLNB in SentiOMIT or omission of ALND in SentiMACRO
- patients with </=2 macrometastasis and omission of ALND (Experimental): breast cancer patients with 1-2 macrometastasis on SLNB and had omission of ALND
  Interventions: Procedure: omission of SLNB in SentiOMIT or omission of ALND in SentiMACRO
- patients with cT1-2N0 and SLNB (No Intervention): early breast cancer patients with cT1-2N0 Luminal A subtype and SLNB
- patients with </=2 macrometastasis and ALND (No Intervention): breast cancer patients with 1-2 macrometastasis on SLNB and had ALND

INTERVENTIONS:
Procedure: omission of SLNB in SentiOMIT or omission of ALND in SentiMACRO — Omission of SLNB in cT1-2N0 or Omission of ALND in patients with </= 2 macrometastasis in SLNB
  Arms: patients with </=2 macrometastasis and omission of ALND; patients with omission of SLNB

SUMMARY:
The treatment and prognosis of breast cancer (BC) are dependent on its molecular subtype and nodal burden. In early BCs with favourable molecular subtype, the incidence of axillary node involvement is low. However, these patients are still subjected to an axillary operation, which can result in additional cost, operating time and morbidities. Similarly, in patients with limited nodal burden of 1-2 metastatic nodes, there is emerging evidence that these patients may need sentinel lymph node biopsy (SLNB) only, instead of an axillary clearance (AC), which has more surgical morbidities.

We aimed to determine if axillary surgery could be safely tailored in BC patients based on their molecular subtype and nodal burden, without compromising their oncological outcomes. This could in turn reduce the morbidities associated with the axillary surgery,

Total 350 patients will be enrolled. 50 patients with early BC and favourable molecular subtype will be enrolled in a pilot study A (SentiOMIT), whereby SLNB is omitted. For eligible patients who declined study A and other stage I-II patients, with preoperative N0 status, undergoing upfront surgery but did not meet the inclusion criteria of Study A, these patients will be enrolled into study B (SentiMACRO) to undergo SLNB.

In study B, the patients will be categorized based on SLNB into 3 groups with 100 patients in each arm: B1 with pN0, B2- 1-2 metastatic nodes and B3- >/=3 metastatic nodes. In Study B, we aim to investigate if the B2 group (100 patients) can be treated with a less invasive procedure of SLNB alone instead of AC, without affecting oncological outcomes. B1 and B3 are controls.

The outcomes for study A and B include short term outcomes such as morbidity rates, cost and operating time savings. Long term outcomes include recurrence and survival rates. This study will allow individualisation of axillary surgery based on the patient's molecular subtype and nodal burden, to benefit patients' care.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged >/=55 years old
* unifocal cancer on imaging
* breast tumour size based on imaging of </=3cm
* no evidence of axillary adenopathy on imaging
* patients with strongly positive ER and PR and negative HER2 on biopsy
* grade 1-2 tumour on core biopsy
* patient who opt for mastectomy

Exclusion Criteria:

* patients with T3/T4 or stage IV disease, patients with preoperative known N+ disease, bilateral breast cancers, patients planned for neoadjuvant chemotherapy, patients with other malignancies.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer
Enrollment: 350 (Estimated)
Dates: Start 2024-02-06 (Estimated); Primary Completion 2033-02-28 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
short term outcomes | from date of surgery, assessed up to 6 months after operation
  complications
short term outcomes | from date of surgery, assessed up to 1 months after operation
  pain score
short term outcomes | from date of surgery, assessed up to 1 months after operation
  cost
long term outcomes | from date of surgery, assessed up to 5 years after operation
  axillary recurrence
long term outcomes | from date of surgery, assessed up to 5 years after operation
  survival

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No